CLINICAL TRIAL: NCT03809000
Title: STEEL: A Randomized Phase II Trial of Salvage Radiotherapy With Standard vs Enhanced Androgen Deprivation Therapy (With Enzalutamide) in Patients With Post-Prostatectomy PSA Recurrences With Aggressive Disease Features
Brief Title: A Study of Salvage Radiotherapy With or Without Enzalutamide in Recurrent Prostate Cancer Following Surgery
Acronym: STEEL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RTOG Foundation, Inc. (Other)
Collaborators: Pfizer (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 3506; STEEL (Other: RTOG Foundation)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Post-prostatectomy; Enzalutamide; STEEL
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Image-Guided; enzalutamide; bicalutamide; Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; luprolide acetate gel depot; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salvage Radiation Therapy (SRT) + Standard androgen deprivation therapy (ADT) (Active Comparator): Standard ADT: 24 months of GnRH analog (any formulation) with optional 1-4 months of bicalutamide (50 mg/day).
  SRT: Starting within 0-70 days of initiation of GnRH analog, 66.6-70.2 Gy as 1.8 Gy/fraction in 37-39 fractions or 66.0-70.0 Gy as 2.0 Gy/fraction in 33-35 fractions lasting approximately 7-8 weeks, and optional lymph node boost.
  Interventions: Radiation: Radiation Therapy; Drug: Bicalutamide; Drug: GnRH analog
- Salvage Radiation Therapy + Enhanced ADT (Experimental): Enhanced ADT: 24 months of GnRH analog (any formulation) with 24 months of enzalutamide (160 mg/day).
  SRT: Starting within 0-70 days of initiation of GnRH analog, 66.6-70.2 Gy as 1.8 Gy/fraction in 37-39 fractions or 66.0-70.0 Gy as 2.0 Gy/fraction in 33-35 fractions lasting approximately 7-8 weeks, and optional lymph node boost.
  Interventions: Radiation: Radiation Therapy; Drug: Enzalutamide; Drug: GnRH analog

INTERVENTIONS:
Radiation: Radiation Therapy — daily fractions
  Other Names: RT; Image-Guided Radiation Therapy (IGRT); Radiotherapy
Drug: Enzalutamide — tablet
  Other Names: Xtandi®
  Arms: Salvage Radiation Therapy + Enhanced ADT
Drug: Bicalutamide — tablet
  Other Names: Casodex®
  Arms: Salvage Radiation Therapy (SRT) + Standard androgen deprivation therapy (ADT)
Drug: GnRH analog — Injection
  Other Names: Gonadotropin-releasing hormone analog; Lupron®; leuprolide acetate; goserelin acetate; Eligard™; Viadur™; Zoladex®; Trelstar®

SUMMARY:
Patients with post-prostatectomy PSA (Prostate Specific Antigen) recurrences with aggressive disease features will receive salvage radiation therapy and standard androgen deprivation therapy (ADT) or enhanced ADT to determine if there is any improvement in progression-free survival when enhanced ADT is used compared to standard ADT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine whether, in men with post-prostatectomy PSA (prostate specific antigen) recurrences with aggressive disease features, salvage radiotherapy (SRT) with enhanced androgen deprivation therapy (ADT), consisting of enzalutamide (MDV3100) and a GnRH analog, will improve progression-free survival compared to SRT with standard GnRH analog -based ADT.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven adenocarcinoma confirmed by prostatectomy performed within 10 years prior to registration and any type of radical prostatectomy is permitted, including retropubic, perineal, laparoscopic or robotically assisted.
* Prostate-specific antigen (PSA) level (≥ 0.2 ng/mL) within 120 days prior to registration. Patients must have a PSA ≥ 0.2 ng/mL prior to starting ADT. For patients being followed by an ultrasensitive PSA assay, a serum PSA concentration of ≥ 0.10 ng/mL will be considered eligible.
* GnRH analog may be started no more than 42 days prior study entry.
* Hemoglobin ≥ 9.0 g/dL, independent of transfusion and/or growth factors within 90 days prior to registration.
* Platelet count ≥ 75,000 x 10^9/µL independent of transfusion and/or growth factors within 90 days prior to registration.
* At least 1 of the following aggressive features:

  * Gleason score of 8-10 (note any Gleason score is eligible)
  * Seminal vesicle invasion (SVI) (note any pT stage American Joint Committee on Cancer (AJCC) v8.0 is eligible but a pT stage

    ≥ pT3b is considered aggressive)
  * Locoregional node involvement at radical prostatectomy (RP) (pN1)
  * Persistently elevated PSA post-RP nadir (PEPP) defined as PSA > 0.1 ng/mL after radical prostatectomy
  * PSA ≥ 0.7 ng/mL
* Serum albumin ≥ 3.0 g/dL within 90 days prior to registration
* Glomerular filtration rate (GFR) ≥35 mL/min estimated by Cockcroft-Gault or measured directly by 24 hour urine creatinine within 90 days prior to registration.
* Serum total bilirubin ≤1.5 × upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, subject is eligible) within 90 days prior to registration.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5 × ULN within 90 days prior to registration.
* History and physical with Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 or within 90 days prior to registration.

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease with the exception of locoregional lymph nodes.
* Prior invasive malignancy (except non-melanomatous skin cancer carcinoma in situ of the male breast, penis, oral cavity, or stage Ta of the bladder, or stage I completely resected melanoma) unless disease free for a minimum of 2 years).
* Prior systemic chemotherapy for the study cancer. Note: prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* History of any of the following:

  * Documented inflammatory bowel disease
  * Transmural myocardial infarction within the last 4 months prior to registration.
  * New York Heart Association Functional Classification III/IV within 4 months prior to registration.
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 4 months prior to registration
  * History of loss of consciousness or transient ischemic attack within 12 months prior to randomization
  * History of seizure disorder or condition that may predispose to seizure (e.g. prior cortical stroke or significant brain trauma)
  * History of uncontrolled hypertension defined as a sustained systolic blood pressure in excess of 150 mmHg or a sustained diastolic blood pressure in excess of 90 mmHg despite optimized antihypertensive therapy.
  * History of repeated falls and fractures over the past 12 months that in the opinion of the treating investigator would put the patient at risk for poor bone outcomes from androgen receptor targeted therapy
* Known gastrointestinal disorder affecting absorption of oral medications.
* Active uncontrolled infection defined as an identified infectious condition that requires active therapy that has not yet been completed.
* HIV positive patients with CD4 count < 200 cells/microliter within 30 days prior to registration OR HIV patients under treatment with highly active antiretroviral therapy (HAART) within 30 days prior to registration regardless of CD4 count. Note: HIV testing is not required for eligibility for this protocol as it is self-reported. This exclusion criterion is necessary because the treatments involved in this protocol may be immunosuppressive and/or interact with HAART.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2029-09-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD, Principal Investigator — RTOG Foundation; Hiram Gay, MD, Principal Investigator — RTOG Foundation
Locations (108):
- United States (106):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale East, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Scottsdale North, Scottsdale, Arizona
  - Arizona Center for Cancer Care - Surprise, Surprise, Arizona
  - Marin Cancer Care, Inc., Greenbrae, California
  - Marin Health Medical Center, Greenbrae, California
  - University of Southern California, Los Angeles, California
  - USC Medical Center - Los Angeles County, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Roseville Radiation Oncology Center, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - University of Florida Health Science Center, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Nancy N. & J.C. Lewis Cancer & Research Pavilion, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Kansas University Cancer Center Overland Park, Overland Park, Kansas
  - Kansas University Cancer Center Westwood, Westwood, Kansas
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network/Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Coastal Cancer Treatment Center - Bath, Bath, Maine
  - Waldo Count General Hospital - Belfast, Belfast, Maine
  - Maine Health/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Maine Health/Stephens Memorial - Norway, Norway, Maine
  - Maine Medical Center - Bramhall S Portland, Portland, Maine
  - Penobscot Bay Medical Center - Rockport, Rockport, Maine
  - Maine Health CC of York County - Sanford, Sanford, Maine
  - Maine Health/SMHCancer Care and Blood Disorders - Sanford, Sanford, Maine
  - Maine Medical Cancer Center - Scarborough Campus, Scarborough, Maine
  - Maine Medical Partners - South Portland, South Portland, Maine
  - McLaren Cancer Institute - Bloomfield, Bloomfield, Michigan
  - 21st Century Oncology MHP - Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute - Clarkston, Clarkston, Michigan
  - William Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State/Karmanos Cancer Institute, Detroit, Michigan
  - 21st Century Oncology MHP - Farmington, Farmington Hills, Michigan
  - McLaren Cancer Institute - Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - McLaren Cancer Institute - Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians - Lansing, Lansing, Michigan
  - McLaren Cancer Institute - Lapeer Region, Lapeer, Michigan
  - 21st Century Oncology MHP - Macomb, Macomb, Michigan
  - 21st Century Oncology MHP - Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute - Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute - Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute - Owosso, Owosso, Michigan
  - McLaren Cancer Institute - Northern Michigan, Petoskey, Michigan
  - McLaren Cancer Institute - Port Huron, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Sterling Heights, Michigan
  - 21st Century Oncology MHP - Troy, Troy, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA - Maplewood, Maplewood, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - HealthPartners, Inc., Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Kansas University Cancer Center North, Kansas City, Missouri
  - Kansas University Cancer Center Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University Physicians at Oneida, Oneida, New York
  - Upstate Cancer Center Radiation Oncology at Oneida, Oneida, New York
  - University Physicians at Oswego, Oswego, New York
  - Upstate Cancer Radiation Oncology at Oswego, Oswego, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - UNC Rex Cancer Center, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - WellSpan Health - Ephrata Cancer Center, Ephrata, Pennsylvania
  - WellSpan Health - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - WellSpan Health - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - University of Pittsburgh Medical Center - Shadyside Hospital, Pittsburgh, Pennsylvania
  - WellSpan Health - York Hospital, York, Pennsylvania
  - Gibbs Cancer Center - Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - UT Southwestern/Simmons Cancer Center - Dallas, Dallas, Texas
  - American Fork Hospital, American Fork, Utah
  - Cedar City Hospital, Cedar City, Utah
  - Logan Regional Medical Center, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Dartmouth Hitchcock Medical Center/Norris Cancer Ctr. - St. Johnsbury, Saint Johnsbury, Vermont
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Aspirus Langlade Hospital, Antigo, Wisconsin
  - University Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square, Oak Creek, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (2):
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSS de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Salvage Radiation Therapy (SRT) + Standard Androgen Deprivation Therapy (ADT): Standard ADT: 24 months of gonadotropin-releasing hormone (GnRH) analog (any formulation) with optional 1-4 months of bicalutamide (50 mg/day).
  SRT: Starting within 0-70 days of initiation of GnRH analog, 66.6-70.2 Gy as 1.8 Gy/fraction in 37-39 fractions or 66.0-70.0 Gy as 2.0 Gy/fraction in 33-35 fractions lasting approximately 7-8 weeks, and optional lymph node boost.
Period: Overall Study
Arm/Group | Salvage Radiation Therapy (SRT) + Standard Androgen Deprivation Therapy (ADT) | Salvage Radiation Therapy + Enhanced ADT
Started | 98 | 90
Adverse Event Population (Randomized participants who started treatment and were assessed for adverse events.) | 98 | 89
Completed (Participants contributing data to results are considered to have completed the study.) | 98 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- SRT + Standard ADT: Standard ADT: 24 months of GnRH analog (any formulation) with optional 1-4 months of bicalutamide (50 mg/day).
  SRT: Starting within 0-70 days of initiation of GnRH analog, 66.6-70.2 Gy as 1.8 Gy/fraction in 37-39 fractions or 66.0-70.0 Gy as 2.0 Gy/fraction in 33-35 fractions lasting approximately 7-8 weeks, and optional lymph node boost.
- SRT + Enhanced ADT: Enhanced ADT: 24 months of GnRH analog (any formulation) with 24 months of enzalutamide (160 mg/day).
  SRT: Starting within 0-70 days of initiation of GnRH analog, 66.6-70.2 Gy as 1.8 Gy/fraction in 37-39 fractions or 66.0-70.0 Gy as 2.0 Gy/fraction in 33-35 fractions lasting approximately 7-8 weeks, and optional lymph node boost.
- Total: Total of all reporting groups
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT | Total
Number analyzed (Participants) | 98 | 90 | 188
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 78] | 63 [47 to 77] | 64 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 98 | 90 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 89 | 82 | 171
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 15 | 21
  White | 85 | 67 | 152
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 5 | 2 | 7
Baseline PSA [Median (Full Range); unit: ng/mL] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  ng/mL | 0.565 [0.11 to 9.56] | 0.785 [0.109 to 24.8] | 0.605 [0.109 to 24.8]
Pathologic T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 8th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b. Higher numbers and/or letters indicate worse condition.
  Participants
    T2 | 21 | 15 | 36
    T3 | 2 | 2 | 4
    T3a | 31 | 28 | 59
    T3b | 42 | 43 | 85
    T4 | 2 | 2 | 4
Pathologic N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 8th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants
    N0 | 63 | 63 | 126
    N1 | 20 | 21 | 41
    NX | 15 | 6 | 21
Gleason Score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    6 | 1 | 0 | 1
    7 | 39 | 34 | 73
    8 | 11 | 5 | 16
    9 | 46 | 51 | 97
    10 | 1 | 0 | 1
ECOG (Eastern Cooperative Oncology Group) Performance Status Scale [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death. (Only 0 and 1 were allowed for this study.)
  Participants
    0 | 90 | 77 | 167
    1 | 8 | 13 | 21
Number of aggressive features [Count of Participants; unit: Participants] — The following are considered aggressive features:
  * Gleason score of 8-10 (note any Gleason score is eligible)
  * Seminal vesicle invasion (SVI) (note any pT stage is eligible [AJCC v8.0] but pT stage ≥ pT3b is considered aggressive)
  * Locoregional node involvement (pN1) at radical prostatectomy (RP)
  * Persistently elevated PSA post-RP (PEPP) defined as PSA > 0.1 ng/mL after radical prostatectomy
  * PSA ≥0.7 ng/mL
  Participants
    1 | 30 | 23 | 53
    > 1 | 68 | 67 | 135

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive Without Progression (Progression-Free Survival)
Description: Progression-free survival (PFS) is estimated by the Kaplan-Meier method. PFS time is measured from randomization to the date of first PFS failure (biochemical or clinical failure, initiation of new unplanned anticancer treatment, or death from any cause) or last known follow-up (censored). Analysis was to occur after progression or death was reported for 101 participants. Biochemical failure is defined as first post-RT detectable PSA (PSA ≥ 0.05). Clinical failure is defined as either a local, regional, or distant failure.
Time Frame: From randomization to first failure or last known follow-up. Median follow-up time at the time of analysis was 33.1 months. The 1- and 2-year estimates are reported.
Population: Randomized participants
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
percentage of participants
  1 year | 38.3 [32.0 to 44.7] | 45.5 [38.6 to 52.4]
  2 years | 32.1 [26.0 to 38.2] | 38.3 [31.5 to 45.0]
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; After protocol amendments, the 3-year PFS rate of the standard arm was expected to be 24%. Assuming a hazard ratio of 0.65 (treatment/control) results in a hypothesized 3-year PFS rate of 39.5% on the enhanced ADT arm. A one-sided log-rank test with alpha=0.10 at 80% statistical power was calculated to require 101 events from 170 patients, taking into account expected accrual rate and follow-up time; Test type: Superiority; p = 0.0671, Log Rank; One-sided significance level = 0.10; Hazard Ratio (HR) = 0.76, 80% CI 2-sided [0.61 to 0.96] — Reference level = standard ADT

2. Secondary Outcome: Percentage of Participants With Biochemical Failure
Description: Biochemical failure is defined as the first detectable post-RT prostate-specific antigen (PSA) value (≥ 0.05) or the initiation of salvage hormone therapy. Failure rates are estimated using the cumulative incidence method, treating death as a competing risk, and otherwise censoring participants alive at time of analysis.
Time Frame: From randomization to first failure, competing event, or last known follow-up, whichever occurs first. Median follow-up time at the time of analysis was 33.1 months. The 1- and 2-year estimates are reported.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
percentage of participants
  1 year | 61.7 [51.1 to 70.6] | 54.6 [43.4 to 64.5]
  2 years | 67.9 [57.5 to 76.3] | 60.6 [49.3 to 70.2]
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.1160, Gray's; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.07] — Reference level = SRT + Standard ADT

3. Secondary Outcome: Percentage of Participants With Alternative Biochemical Failure
Description: Alternative biochemical failure is defined as first post-RT PSA ≥ 0.1 ng/mL or initiation of salvage hormone therapy. Failure rates are estimated using the cumulative incidence method, treating death as a competing risk, and otherwise censoring participants alive at time of analysis.
Time Frame: as for outcome 2
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
percentage of participants
  1 year | 35.9 [26.5 to 45.5] | 31.4 [21.9 to 41.3]
  2 years | 45.4 [35.2 to 55.0] | 39.9 [29.4 to 50.2]
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.1618, Gray's; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.50 to 1.12] — Reference level = SRT + Standard ADT

4. Secondary Outcome: Percentage of Participants With Hormone-refractory Disease
Description: Hormone-refractory disease is defined as three rises in PSA during salvage androgen deprivation, with the date determined as the midway date between the last non-rising PSA and the first of the three rises. Failure rates were to be estimated using the cumulative incidence method, treating death as a competing risk, and otherwise censoring participants alive at time of analysis, but for endpoints with < 10 events overall, such as this one, only the counts of participants with the event are provided.
Time Frame: From randomization to first failure, competing event, or last known follow-up, whichever occurs first. Median follow-up time at the time of analysis was 33.1 months.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
Participants | 0 | 0

5. Secondary Outcome: Percentage of Participants With Distant Metastasis
Description: Distant failure is defined as first radiographic evidence of distant metastasis (e.g., bone scan, computed tomography (CT), magnetic resonance imaging (MRI)). Failure rates were to be estimated using the cumulative incidence method, treating death as a competing risk, and otherwise censoring participants alive at time of analysis, but for endpoints with < 10 events overall, such as this one, only the counts of participants with the event are provided.
Time Frame: as for outcome 4
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
Participants | 6 | 1

6. Secondary Outcome: Percentage of Participants With Prostate Cancer Death
Description: Cause-specific mortality is defined as death due to prostate cancer. Failure rates were to be estimated using the cumulative incidence method, treating death as a competing risk, and otherwise censoring participants alive at time of analysis, but for endpoints with < 10 events overall, such as this one, only the counts of participants with the event are provided.
Time Frame: as for outcome 4
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
Participants | 0 | 0

7. Secondary Outcome: Percentage of Participants Alive (Overall Survival)
Description: Survival rates were to be estimated using the Kaplan-Meier method, censoring participants alive at time of analysis, but for endpoints with < 10 events overall, such as this one, only counts are provided. In this case, the number of participants without event (death), which is the number of participants alive.
Time Frame: From randomization to death or last known follow-up, whichever occurs first. Median follow-up time at the time of analysis was 33.1 months.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
Participants | 96 | 90

8. Secondary Outcome: Change From Baseline to End of RT in the 5-level European Quality of Life Questionnaire (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a self-assessment questionnaire. The index score is computed from 5 items (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each with 5 problem levels (1-none to 5-extreme). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). Change score was calculated by subtracting baseline from later score, with a positive change score indicating improvement.
Time Frame: Baseline and end of radiation treatment (RT). End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality of life study component and who have baseline and end of RT data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 77 | 67
score on a scale | 0.0 (0.1) | 0.0 (0.1)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.7184, t-test, 2 sided

9. Secondary Outcome: Change From Baseline to One Year After End of RT in the EQ-5D-5L Index Score
Description: as for outcome 8
Time Frame: Baseline and one year after end RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality of life study component and who have baseline and one year after end of RT data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 71 | 64
score on a scale | 0.0 (0.1) | 0.0 (0.1)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.5934, t-test, 2 sided

10. Secondary Outcome: Change From Baseline to Two Years After End of RT in the EQ-5D-5L Index Score
Description: as for outcome 8
Time Frame: Baseline and two years after end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality of life study component and who have baseline and two year after end of RT data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 64 | 62
score on a scale | 0.0 (0.1) | 0.0 (0.1)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.7129, t-test, 2 sided

11. Secondary Outcome: Change From Baseline to End of RT in the 7-item Patient Reported Outcomes Measurement Information System - Fatigue Short Form (PROMIS-F SF 7a) [PROMIS Fatigue Score]
Description: The PROMIS fatigue score measures self-reported fatigue symptoms over the past 7 days. Possible raw scores range from 29.4 to 83.2 (higher raw score indicating greater fatigue) and are converted into standardized T-scores (mean=50, standard deviation=10) with higher scores also indicating greater fatigue. Change score is calculated by subtracting baseline T-score from later T-score, with a positive change score indicating increased fatigue.
Time Frame: Baseline and end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality of life study component and who have baseline and end of RT data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 74 | 64
score on a scale | 3.4 (7.8) | 6.8 (6.4)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.006258, t-test, 2 sided

12. Secondary Outcome: Change From Baseline to One Year After the End of RT in the 7-item Patient Reported Outcomes Measurement Information System - Fatigue Short Form (PROMIS-F SF 7a) [PROMIS Fatigue Score]
Description: as for outcome 11
Time Frame: Baseline and one year after end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality of life study component and who have baseline and end of RT data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 72 | 61
score on a scale | 4.0 (7.4) | 7.0 (8.0)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.0263, t-test, 2 sided

13. Secondary Outcome: Change From Baseline to Two Years After the End of RT in the 7-item Patient Reported Outcomes Measurement Information System - Fatigue Short Form (PROMIS-F SF 7a) [PROMIS Fatigue Score]
Description: as for outcome 11
Time Frame: Baseline, two years after end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who consented to the quality-of-life study component and who have baseline and two years after end of RT data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 66 | 60
score on a scale | 4.0 (7.5) | 5.0 (7.8)
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.4599, t-test, 2 sided

14. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported CTCAE v5
Description: Common Terminology Criteria for Adverse Events (version 5) grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to death or last known follow-up. Median follow-up time at the time of analysis was 33.1 months.
Population: Randomized participants who started protocol treatment and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 89
Participants
  None | 8 | 3
  Grade 1 | 19 | 9
  Grade 2 | 38 | 32
  Grade 3 | 27 | 39
  Grade 4 | 6 | 6
  Grade 5 | 0 | 0

15. Secondary Outcome: Number of Participants Any Adverse Event Occuring Within 30 Days Following the End of Treatment
Description: as for outcome 14
Time Frame: From randomization to 30 days after the end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who started protocol treatment and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 89
Participants | 86 | 83
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.3138, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.62 to 4.41] — Reference level = SRT + Standard ADT

16. Secondary Outcome: Number of Participants With Any Grade 3+ Adverse Event Occuring After 30 Days Following the End of RT
Description: as for outcome 14
Time Frame: From 31 days after the end of RT to death or last known follow-up. Median follow-up was 33.1 months. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants who started protocol treatment, were assessed for adverse events, and alive 30 days after radiation therapy ended.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 89
Participants | 27 | 30
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.3889, Chi-squared

17. Secondary Outcome: Number of Participants With Post-baseline Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Scores ≥ 3
Description: PRO-CTCAE is a patient-reported outcome (PRO) measurement system developed to evaluate symptomatic toxicity in patients on cancer clinical trials, asking the patient about experience over the last seven days. Scores may reflect worst severity of the symptom (0=None, 1=Mild, 2=Moderate, 3=Severe, and 4=Very severe), frequency of the symptom (0=Never, 1=Rarely, 2=Occasionally, 3=Frequently, 4=Almost constantly), or the symptom's interference with one's "usual or daily activities" (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). The symptom row title will indicate "Severity", "Frequency", or "Interference". All scores are compared between arms; statistical analysis results are entered for p-values < 0.05.
Time Frame: End of RT, one and two years after the end of RT. End of RT can vary greatly depending on when it starts, which can be from 0 to 70 days from the start of ADT, and lasting 7-8 weeks.
Population: Randomized participants with PRO-CTCAE data.
Measure: Count of Participants; unit: Participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 96 | 87
Participants
  Taste Changes Severity | 3 | 8
  Decreased Appetite Severity | 2 | 6
  Decreased Appetite Interference | 2 | 4
  Nausea Frequency | 8 | 8
  Nausea Severity | 7 | 3
  Constipation Severity | 13 | 9
  Loose Stool Frequency | 30 | 19
  Abdominal Pain Frequency | 19 | 14
  Abdominal Pain Severity | 13 | 9
  Abdominal Pain Interference | 10 | 7
  Bowel Movement Control Frequency | 9 | 5
  Bowel Movement Control Interference | 7 | 5
  Racing Heartbeat Frequency | 5 | 6
  Racing Heartbeat Severity | 3 | 1
  Itchy Skin Severity | 10 | 3
  Concentration Problems Severity | 9 | 11
  Concentration Problems Interference | 12 | 11
  Memory Problems Severity | 7 | 11
  Memory Problems Interference | 8 | 11
  Headache Frequency | 12 | 9
  Headache Severity | 5 | 9
  Headache Interference | 5 | 6
  Fatigue Severity | 29 | 31
  Fatigue Interference | 31 | 34
  Pain with Urination Severity | 4 | 6
  Urinary Urgency Frequency | 38 | 37
  Urinary Urgency Interference | 23 | 25
  Frequent Urination Frequency | 46 | 45
  Frequent Urination Interference | 25 | 24
  Urine Control Loss Frequency | 39 | 39
  Urine Control Loss Interference | 22 | 28
  Erection Difficulty Severity: number analyzed (Participants) | 96 | 86
  Erection Difficulty Severity | 40 | 24
  Ejaculation Problems Frequency | 26 | 18
  Decreased Sexual Interest Severity | 42 | 33
  Breast Tenderness Severity | 7 | 7
  Hot Flashes Frequency | 56 | 63
  Hot Flashes Severity | 32 | 44
  Pain Frequency | 35 | 33
  Pain Severity | 21 | 23
  Pain Interference | 16 | 23
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Hot Flashes Frequency; Test type: Superiority; p = 0.0461, t-test, 2 sided
Statistical Analysis 2: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Hot Flashes Severity; Test type: Superiority; p = 0.0181, t-test, 2 sided

18. Post Hoc Outcome: Percentage of Participants Alive Without Progression (Progression-Free Survival) [Alternate Definition]
Description: Progression-free survival (PFS) is estimated by the Kaplan-Meier method. PFS time is measured from randomization to the date of first PFS failure (biochemical or clinical failure, initiation of new unplanned anticancer treatment, or death from any cause) or last known follow-up (censored). Analysis was to occur after progression or death was reported for 101 participants. Biochemical failure is defined as first post-RT PSA ≥ 0.2. Clinical failure is defined as either a local, regional, or distant failure.
Time Frame: From randomization to first failure or last known follow-up. Medium follow-up time at the time of analysis was 33.1 months. The 1- and 2-year estimates are reported.
Population: Randomized participants
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
Number analyzed (Participants) | 98 | 90
percentage of participants
  1 year | 87.5 [83.2 to 91.8] | 91.9 [88.1 to 95.6]
  2 years | 78.8 [73.4 to 84.2] | 88.3 [83.8 to 92.7]
Statistical Analysis 1: Comparison: SRT + Standard ADT vs SRT + Enhanced ADT; Test type: Superiority; p = 0.10, Log Rank — one-sided p-value; Hazard Ratio (HR) = 0.62, 80% CI 2-sided [0.42 to 0.91]

ADVERSE EVENTS:
Time Frame: Baseline to the date of last known follow-up. Maximum follow-up time was 40.1 months.
Description: All-cause mortality was assessed in randomized participants. Adverse events were assessed in randomized participants who started protocol treatment and were assessed for adverse events.
Arm/Group | SRT + Standard ADT | SRT + Enhanced ADT
All-Cause Mortality (participants affected / at risk) | 2/98 | 0/90
Serious Adverse Events (participants affected / at risk) | 11/98 | 17/89
Other Adverse Events (participants affected / at risk) | 89/98 | 87/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRT + Standard ADT (N=98) | SRT + Enhanced ADT (N=89)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Eye disorders - Other (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Localized edema (General disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Lymph gland infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Salivary gland infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Creatinine increased (Investigations) | 0 | 1
Investigations - Other (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Movements involuntary (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 3
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thromboembolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRT + Standard ADT (N=98) | SRT + Enhanced ADT (N=89)
Anemia (Blood and lymphatic system disorders) | 16 | 33
Blurred vision (Eye disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 13 | 15
Constipation (Gastrointestinal disorders) | 28 | 25
Diarrhea (Gastrointestinal disorders) | 61 | 48
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 12 | 12
Nausea (Gastrointestinal disorders) | 18 | 28
Proctitis (Gastrointestinal disorders) | 9 | 7
Rectal hemorrhage (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 8 | 6
Edema limbs (General disorders) | 4 | 8
Fatigue (General disorders) | 70 | 65
Non-cardiac chest pain (General disorders) | 5 | 2
Pain (General disorders) | 10 | 7
Infections and infestations - Other (Infections and infestations) | 6 | 11
Urinary tract infection (Infections and infestations) | 6 | 3
Fall (Injury, poisoning and procedural complications) | 7 | 8
Alanine aminotransferase increased (Investigations) | 2 | 13
Aspartate aminotransferase increased (Investigations) | 1 | 12
Creatinine increased (Investigations) | 7 | 8
Investigations - Other (Investigations) | 4 | 5
Lymphocyte count decreased (Investigations) | 13 | 25
Neutrophil count decreased (Investigations) | 2 | 9
Platelet count decreased (Investigations) | 5 | 9
Weight gain (Investigations) | 16 | 16
Weight loss (Investigations) | 5 | 10
White blood cell decreased (Investigations) | 12 | 18
Anorexia (Metabolism and nutrition disorders) | 6 | 14
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 18
Hypokalemia (Metabolism and nutrition disorders) | 6 | 6
Hyponatremia (Metabolism and nutrition disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 17
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 | 13
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 9 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9
Concentration impairment (Nervous system disorders) | 5 | 9
Dizziness (Nervous system disorders) | 9 | 16
Dysgeusia (Nervous system disorders) | 4 | 11
Extrapyramidal disorder (Nervous system disorders) | 0 | 5
Headache (Nervous system disorders) | 16 | 16
Memory impairment (Nervous system disorders) | 7 | 16
Paresthesia (Nervous system disorders) | 3 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 5
Anxiety (Psychiatric disorders) | 5 | 5
Confusion (Psychiatric disorders) | 1 | 5
Depression (Psychiatric disorders) | 13 | 8
Insomnia (Psychiatric disorders) | 9 | 17
Libido decreased (Psychiatric disorders) | 11 | 12
Cystitis noninfective (Renal and urinary disorders) | 12 | 8
Dysuria (Renal and urinary disorders) | 21 | 18
Hematuria (Renal and urinary disorders) | 25 | 17
Renal and urinary disorders - Other (Renal and urinary disorders) | 13 | 13
Urinary frequency (Renal and urinary disorders) | 39 | 35
Urinary incontinence (Renal and urinary disorders) | 43 | 30
Urinary retention (Renal and urinary disorders) | 14 | 4
Urinary tract obstruction (Renal and urinary disorders) | 5 | 5
Urinary urgency (Renal and urinary disorders) | 36 | 25
Erectile dysfunction (Reproductive system and breast disorders) | 17 | 9
Gynecomastia (Reproductive system and breast disorders) | 14 | 10
Pelvic pain (Reproductive system and breast disorders) | 5 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 6
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 8 | 11
Hot flashes (Vascular disorders) | 72 | 73
Hypertension (Vascular disorders) | 25 | 28

LIMITATIONS AND CAVEATS:
The sample size calculation was modified due to a change in eligibility, however the sample size itself remained the same at 242 patients since the hazard ratio was reduced of 0.65 to 0.63. Later, a change in the definition of biochemical failure which is a component of the primary endpoint of PFS decreased the sample size to 170 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03809000/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03809000/ICF_001.pdf